CLINICAL TRIAL: NCT02856477
Title: Pharmacogenetic in the Therapeutic Strategy in Depressed Elderly
Brief Title: Pharmacogenetic and Antidepressant Treatment in Elderly
Acronym: Pharmacogeneti
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: R/2007/32
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Urinalysis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- adapted treatment (Experimental): the treatment dose is adapted to the metabolic capacity of the patient. intervention: urine analysis
  Interventions: Biological: urine analysis
- non-adaptated treatment (Experimental): the treatment dose is adapted to the metabolic capacity of the patient. intervention: urine analysis
  Interventions: Biological: urine analysis

INTERVENTIONS:
Biological: urine analysis — a sample of urine is collected during 8 hours.

SUMMARY:
The study aims to assess the therapeutic benefits of the adaptation of the antidepressant dose to the metabolic capacity (cytochrome P450 2D6) of elderly depressed patients.

Therapeutic benefits are evaluated through the enhancement of efficiency, decrease of the action time and the after effects.

ELIGIBILITY:
Inclusion Criteria:

* current major depressive disorder
* antidepressant treatment

Exclusion Criteria:

* dextromethorphan contra-indication
* other psychiatric disorder
* kidney failure
* liver failure mini mental State Examination (MMSE)<18

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
patient remission | 6 months
  remission is defined by a Montgomery and asberg depression rating (MADRS) score<10.

CONTACTS AND LOCATIONS:
Overall Officials: pierre Vandel, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHU Besancon, Besançon, Doubs, France

IPD SHARING:
Plan to Share IPD: No